CLINICAL TRIAL: NCT03649243
Title: Propolis as Adjuvant in the Healing of Human Diabetic Foot Wounds Receiving Care in Diagnostic and Treatment Center From Regional Hospital of Talca
Brief Title: Propolis as Adjuvant in the Healing of Human Diabetic Foot Wounds
Status: Completed | Type: Observational
Sponsor: University of Talca (Other)
Collaborators: Hospital Regional de Talca (Unknown)
Responsible Party: Principal Investigator, Jessica Zuñiga-Hernandez, Head Laboratory, Unidad de Farmacología, Laboratorio de Investigaciones Médicas, Escuela de Medicina,, University of Talca
Other Study IDs: 2015-c03
Record Dates: First submitted 2018-06-12; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Foot wounds; oxidative stress; inflammation; propolis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — biopsy of the ulcer site, after debridement
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propolis group: The patients receive propolis (3% in Propylene Glycol) in all the wound surface in each healing until cicatrisation or at least 8 weeks. (n=20)
  Interventions: Drug: Propolis spray
- control group: the patients received the same care in the healing of their wounds, but no new component or propolis 3% was administered (n=8)

INTERVENTIONS:
Drug: Propolis spray — Propolis was added at the site of injury, 3 puff for any wound in the foot of patients. All the patients decide voluntary if they want to receive the propolis spray treatment or only receive they normal wound healing care.
  Groups: Propolis group

SUMMARY:
The general objective of the project is "To evaluate the effect of the administration of propolis extract as a coadjuvant in the treatment of diabetic foot ulcers in patients receiving cures in the Specialties Polyclinic of the Regional Hospital of Talca, Maule Region", which will be used Propolis produced in the area, (Laboratorios Rotterdam Ltda.) used in topical form.

It has been described that among the benefits produced by Propolis, is its anti-inflammatory, antioxidant effect and that the topical application of it is well tolerated, improving the healing of human diabetic foot ulcer.

DETAILED DESCRIPTION:
They will be invited to enter the study, at no cost, to 72 patients seen in the Specialty Clinic of the Regional Hospital of Talca, who have a history of diabetic feet with ulcers and who are in treatment with cures and who meet the following criteria. inclusion:

* People with Diabetes Mellitus (DM), older than 18 years, type 1 or 2, with known evolution of their diabetes between 2 and 15 years.
* Carriers of diabetic foot ulcers
* Without other important diseases

Patients who present the following criteria will be excluded from the study:

* Propolis allergy
* Serious circulation problems
* Foot burns
* Psychological conditions, or distances that prevent regular attendance to all required cures.

According to the programmed, 72 people will be admitted to the study, of which half will receive Propolis application on their wound at the end of their usual healing, for a maximum period of 75 days; while the other half will maintain the usual cure without Propolis.

All participants must maintain the usual treatment of their illness, as well as the usual type and frequency of their cures and maintain their physical activity according to the medical indication during this period. After 75 days, those who did not receive Propolis will have the possibility to receive it in the same way for 75 days.

All patients in the study must have a recent basic evaluation of their Diabetes performed in their office or the Specialties Polyclinic of the Regional Hospital of Talca at the beginning (up to 30 days prior) and at the end of the treatment, consisting of glycemia and glycosylated hemoglobin.

Tissue samples will be taken from your wound to make measurements of inflammation, degree of healing, infectionand oxidative stress, at the beginning, week 3, 6 and at the end of the study (75 days). The sample at the end of the study will only be obtained if the wound is still open.

In addition, at the beginning and at the end a blood sample of 5cc will be taken to measure levels of inflammatory markers and oxidative stress in blood.

These samples will be taken in the same Specialty Clinic of the Regional Hospital of Talca, but they will be transferred to be processed in the Clinical Biochemistry Laboratory of the Faculty of Health Sciences and the School of Medicine of the University of Talca. . Samples will be stored frozen at -80 ° C, under a code to guarantee confidentiality, for a period of 2 years, after which they will be eliminated.

During the last care / healing that the nurse does to the patient, you will be asked to complete a survey with questions to collect personal opinions about the effect of topical propolis.

Benefits: It has been described that the topical application of Propolis can improve the healing of human diabetic foot ulcer.

ELIGIBILITY:
Inclusion Criteria:

* DM type 1 or 2 with complicated foot diabetics wounds.
* 18-80 years old

Exclusion Criteria:

* Propolis allergy
* Critical ischemia
* Severe infection
* Psycho-social conditions that avoid regular attendance at health aid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to patients undergoing treatment for diabetic foot in the regional hospital of Talca, are in personalized pharmacological treatment, nursing care for each of the diabetic foot ulcers and control at least 2 times a week for healing.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
allergenic to propolis analysis | through study completion, with an average of 8 months
  All patients were analyzed for the probability of allergenic reaction. It was done on the dermal reaction compared to the reaction to a single dose of histamine.

SECONDARY OUTCOMES:
obtaining biopses | the first biopses was obtained at time zero of enrollment and every 4 weeks, until the wound close or at time 12 weeks (end point of the biopses obtaining)
  obtaining wound biopsies for histological and molecular analysis

CONTACTS AND LOCATIONS:
Overall Officials: elba Leiva, Mg, Study Director — University of Talca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mujica V, Orrego R, Fuentealba R, Leiva E, Zuniga-Hernandez J. Propolis as an Adjuvant in the Healing of Human Diabetic Foot Wounds Receiving Care in the Diagnostic and Treatment Centre from the Regional Hospital of Talca. J Diabetes Res. 2019 Sep 12;2019:2507578. doi: 10.1155/2019/2507578. eCollection 2019. PMID 31612147